CLINICAL TRIAL: NCT03925181
Title: A Recovery-Oriented Counselling Group: Supporting Physical, Emotional, and Social Recovery Processes of Critical Care Patients in the ICU Recovery Clinic
Brief Title: A Recovery-Oriented Counselling Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Tanya Mudry, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REB18-2105
Record Dates: First submitted 2019-04-10; First posted 2019-04-24 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Post-Intensive Care Recovery

STUDY DESIGN:
Intervention Model Description: In total, 12 ICU survivors will be recruited along with their 12 caregivers. Once participants have been recruited, they (and their caregivers) will be randomly assigned to 2 arms: intervention or no intervention (waitlist control). The waitlist control group will receive the intervention in the second arm after the first intervention arm is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Recovery counselling group.
  Interventions: Behavioral: Counselling Group
- Waitlist control (No Intervention): Waitlist control group. Will receive intervention after arm one is complete.

INTERVENTIONS:
Behavioral: Counselling Group — All sessions will be based off of SAMHSA's recovery curriculum but tailored to the participants recovering from the ICU and their caregivers. Throughout the 6-weeks, the sessions will be holistic, strengths-based, hopeful, respectful, relational, and subjective, while emphasizing social relationships, social contexts, and meaning and purpose.
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate a recovery-oriented group counselling program for post-discharged critical illness survivors and their caregivers.

DETAILED DESCRIPTION:
The purpose of this pilot project is to develop and evaluate a recovery-oriented counselling group to support the physical, emotional, and social recovery processes of critical care survivors who access the services of the Calgary ICU Recovery Clinics. Upon discharge, critical care survivors are faced with challenges related to their stay in the Intensive Care Unit (ICU), as well as long-term recovery from critical illness. These challenges impact survivors' physical, emotional, social recovery processes, which reduce quality of life, delay (re)integration into their communities, and cause further health problems. Social support and counselling groups show therapeutic promise in supporting recovery processes by increasing social connection, quality of life, acquisition of skills, and emotional and psychological wellbeing.

The purpose of this study is to evaluate a recovery-oriented group counselling program for post-discharged critical illness survivors and their caregivers. The investigators will utilize Substance Abuse and Mental Health Service Administration's (SAMHSA) evidence-based recovery curriculum to develop a counsellor-facilitated recovery-oriented group for patients and caregivers focusing on peer support, relationships, evidence-based strategies, daily life, purpose and meaning-making, strengths, and resilience.

The research objectives are:

* Implement a recovery-oriented counselling group for ICU Recovery Clinic patients and their caregivers.
* Evaluate the recovery-oriented counselling group as situated within the Calgary ICU Recovery Clinic.

The investigators will utilize a Randomized Controlled Trial (RCT) design (non-clinical trial). Participants will be randomized into a treatment (intervention) or wait-list control group. Participants in the wait-list control group will be offered the intervention after the treatment group has completed the intervention group. The investigators will evaluate the intervention through the use of outcomes measures currently used by the ICU Recovery Clinic in a pre-test (t0), immediate post-test (t1), 3-month (t2), and 6-month (t3) follow-ups. In addition, the investigators will conduct a process evaluation of the intervention via content analysis of audio recorded data from semi-structured interviews and focus groups with participants. Patients and caregivers will participate in separate focus groups.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Spent more than 4 days in the ICU,
* Were discharged into the community within 4 months of transfer out of the ICU (excluding patients who were in hospital long-term)
* Speaks English
* Has a fixed address
* Does not have pre-existing psychiatric diagnoses documented in the ICU transfer summary
* Lives within or surrounding Calgary.

Inclusion Criteria for Caregivers:

* Caregiver of an ICU survivor participant meeting criteria above
* Speaks English
* Has a fixed address
* Lives within or surrounding Calgary.

Exclusion Criteria for Patients:

- Long-term hospital stay

Excluding Criteria for Caregivers:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Impact of Events Scale - Revised (IES-r) | Pre-test, immediately following 6-week group completion, 3-month, and 6-month.
  Change of PTSD symptoms. 22 item questionnaire, each scored 0 to 4 points; Scores higher than 24 are concern for PTSD.
  3 subscales: intrusion subscale (mean range from 0-4), avoidance subscale (mean range from 0-4), hyperarousal subscale (mean range from 0-4).
Patient Health Questionnaire (PHQ-9) | Pre-test, immediately following 6-week group completion, 3-month, and 6-month.
  Change of symptoms of depression. Nine items, each of which is scored 0 to 3 providing a 0-27 severity score with higher values indicating increased severity of depression.
Generalized Anxiety Disorder (GAD-7) | Pre-test, immediately following 6-week group completion, 3-month, and 6-month.
  Change of symptoms of anxiety. Seven items, each of which is scored 0-3 providing a 0-21 severity score with higher value indicating increased severity of anxiety.
Godin Leisure Time Activity Questionnaire | Pre-test, immediately following 6-week group completion, 3-month, and 6-month.
  Change in activity levels. Participant indicates how many times on average they completed exercise (strenuous, moderate, mild) for more than 15-minutes during a typical 7-day period.
Euroqol 5 Dimensions (EQ-5D-5L) | Pre-test, immediately following 6-week group completion, 3-month, and 6-month.
  Change in health status. Participants select their current experience of health on a visual analog scale (VAS) and descriptive system. The descriptive system consists of a 1-5 severity scale (higher values indicating increased severity) for 5 categories of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The VAS records the participant's self-rated health on a vertical, visual analogue scale where the endpoints are labeled "best imaginable health state" and "worst imaginable health state."
Employment questionnaire | Pre-test, immediately following 6-week group completion, 3-month, and 6-month.
  Change of employment status. Participants indicate whether their recent hospital stay has affected their employment by selecting both their current employment status and employment status prior to their hospital stay (i.e. one of the following: employed full-time, employed part-time, unemployed, home-maker, caregiver, student full-time, student part-time, on disability, retired, other).

SECONDARY OUTCOMES:
Focus Group | Immediately following 6-week group completion
  Qualitative semi-structured focus group developed by the researcher to evaluate the program. Topics include: experiences about the group, benefits of the group, examples of changes, and areas of improvement for group development.
Qualitative Survey | Immediately following 6-week group completion
  Qualitative self-report form (not survey or scale) developed by the researcher to on symptomatic changes post-intervention. Questions inquire about: changes in daily activities, fulfillment of roles, social relationships, confidence in coping abilities, changes to routine, participation in leisure activities, hopes for the future, and plans for maintaining recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Mudry, PhD, Principal Investigator — University of Calgary
Locations (1):
- Calgary ICU Recovery Clinic: Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No